CLINICAL TRIAL: NCT01953471
Title: Determination of Minimal Clinically Important Difference of Allergic Rhinitis Symptoms Due to Grass Pollen by the Assessment of the Relationship Between the Symptom Scores and Global Rating of Change Questionnaires on the Quality of Life and Well-being.
Brief Title: Prospective Observational Study for Determination of Minimal Clinically Important Difference of Allergic Rhinitis Symptoms Due to Grass Pollen (Equinoxe 2)
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/09; 2011-A00198-33 (Other: ANSM)
Record Dates: First submitted 2013-09-06; First posted 2013-10-01 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Allergic Rhinitis Due to Grass Pollen
MeSH Terms: interventions — Interleukin-13

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Allergic rhinitis
  Interventions: Other: Allergic rhinitis

INTERVENTIONS:
Other: Allergic rhinitis — Questionnaire

SUMMARY:
Prospective multi-center study carried out in France involving patients with allergic rhinitis. Study in usual care where no specific diagnostic or therapeutic procedure is required. The patients will be asked to fill in Questionnaires on a daily and weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 6 and 65 years.
* Patients who have been informed of the nature and aims of the study and have given their written consent to participate in this study in accordance with local laws and requirements.
* Patient with an Grass pollen-related allergic rhinitis (immunologically and / or symptomatically treated or non treated).
* Patients presented for symptomatic management of allergic rhinitis.
* Patients having Symptoms score ≥ 6.

Exclusion Criteria:

* Patients involved in any other clinical/observational study.
* patients unable to fill in the study questionnaires.
* Patient suffering from any diagnosed disease that may interfere with the evaluation of allergic rhinoconjunctivitis' related quality of life, fatigue and daily activities.
* Patients treated with any drug that may influence the patient's fatigue and/or interfere with psychomotor performance.
* Patients suffering from persistent asthma, or asthma exacerbation during grass pollen season.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with allergic rhinitis due to grass pollen
Sampling Method: Non-Probability Sample
Enrollment: 959 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rhinitis Total Symptoms Score (RTSS), (intensity of each symptom measured on a 4-point scale) compared to a 15-point global rating of change questionnaire. | 6 months per patient

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DEVILLIER, MD, PhD, Principal Investigator — Hôpital Foch
Locations (1):
- Hopital Foch, Suresnes, Île-de-France Region, France